CLINICAL TRIAL: NCT03593031
Title: Functional Neural Mechanism of Vision Therapy for Patients With Convergence Insufficiency
Brief Title: Neural Mechanism of Vision Therapy for Patients With Convergence Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Jersey Institute of Technology (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Dr. Tara Lynn Alvarez, Professor, New Jersey Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F182-13; R01EY023261 (NIH)
Record Dates: First submitted 2018-07-06; First posted 2018-07-19 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Convergence Insufficiency
MeSH Terms: conditions — Ocular Motility Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinician did not know which treatment group. Subjects did not know which treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CI OBVAT (Active Comparator): Patients with Convergence Insufficiency in Active Vision Therapy
  Interventions: Behavioral: Office Based Vergence and Accommodative Therapy
- CI Sham therapy (Sham Comparator): CI Sham therapy
  Interventions: Behavioral: Office Based Vergence and Accommodative Therapy
- Controls OBVAT (Active Comparator): Control receive active therapy
  Interventions: Behavioral: Office Based Vergence and Accommodative Therapy
- Controls Sham (Sham Comparator): Subjects with Normal Binocular Vision will receive a therapy that appears to be therapeutic but does not have any binocular coordination benefits.
  Interventions: Behavioral: Office Based Vergence and Accommodative Therapy

INTERVENTIONS:
Behavioral: Office Based Vergence and Accommodative Therapy — Exercises that will stimulate disparity vergence or accommodation independently and then combined will be used.

SUMMARY:
Convergence insufficiency (CI) is a prevalent binocular vision disorder with symptoms that include double/blurred vision, eyestrain, and headaches when engaged in reading or other near work. CI is present in 4% of the population where approximately 27% of CI patients do not improve even with validated therapy. The project will quantitatively study changes in convergence eye movements and neural substrates before and after validated therapy in CI patients. This knowledge can lead to improvements in currently validated therapy, reduction in therapy sessions, and reduced healthcare costs.

DETAILED DESCRIPTION:
Convergence insufficiency (CI), a prevalent binocular vision disorder in adults and children, is characterized by greater exophoria at near than at distance, reduced fusional convergence amplitude, receded near point of convergence, and a reduced accommodative convergence over accommodation ratio (AC/A). CI is associated with symptoms that include double/blurred vision, eyestrain, and headaches when engaged in reading or other near work, thus interfering with activities of daily living. The recent NEI/NIH multi-center randomized clinical trial, the Convergence Insufficiency Treatment Trial (CITT), demonstrated the effectiveness of Office-Based Vergence and Accommodative Therapy with home reinforcement (OBVAT) for CI, reporting 73% of patients have sustained improvements of vision function and symptoms. The team published the first fMRI neural substrate data evoked using convergence eye movements in CI patients before and then post-OBVAT. The team's results suggest that with the reduction of visual symptoms, the following were observed: 1) an increase in the percent signal change of functional activity in the frontal eye fields, posterior parietal cortex and the cerebellar vermis, 2) an increase in convergence peak velocity, 3) a decrease in the near point of convergence, 4) an increase in positive fusional amplitude and 5) a reduction in the amount of exophoria at near. The aims of the current proposal are to test the following two hypotheses as potential underlying mechanisms of CI that may be improved post OBVAT: 1) a reduced ability to adapt vergence in near and far space via the 'slow' component of vergence and 2) a reduced ability to quickly diminish disparity error via the 'fast' component of vergence. Not only will our quantitative methods integrated with established CITT standards address important questions about potential mechanisms causing CI, this proposal seeks to identify how a validated vergence therapy may remediate symptoms. This proposal will determine whether either of these two potential mechanisms are causing CI by quantifying the following: 1) rate and magnitude of phoria adaptation, 2) forced vergence fixation disparity curves, 3) peak velocity of convergence eye movements (studying visual cues such as disparity, accommodation and proximal stimuli in isolation and combination), and 4) the functional activity of the fast and slow vergence neural substrates prior to, and then after, OBVAT. The assembled study team is particularly knowledgeable in terms of OBVAT, convergence insufficiency, optometry, vision science, oculomotor research, functional imaging, modeling and statistics with the necessary resources to successfully complete both aims of this study. Results from the project's aims can lead to targeted treatments with improved success rates, potentially reducing the time to remediate symptoms, and ultimately reducing health care costs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of symptomatic convergence insufficiency binocularly normal control

Exclusion Criteria:

* history of head trauma any systematic disease that can interfere with vergence or accommodation such as multiple sclerosis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Disparity Vergence Response Amplitude | through study completion, an average of 1 year
  how accurate a patient can fixate on a new target

CONTACTS AND LOCATIONS:
Overall Officials: Atam Dhawan, PhD, Study Director — New Jersey Institute of Technology
Locations (1):
- NJIT, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan in place because the eye movement data collected will be in a proprietary format

REFERENCES:
- [Derived] Fine SN, Rutkowski T, Santos EM, Gohel S, Hajebrahimi F, Scheiman M, Alvarez TL. Heath components of objective accommodative responses for convergence insufficiency participants compared with those with binocularly normal vision. Optom Vis Sci. 2025 Dec 1;102(12):731-742. doi: 10.1097/OPX.0000000000002307. Epub 2025 Nov 18. PMID 41252526
- [Derived] Hajebrahimi F, Sangoi A, Scheiman M, Santos E, Gohel S, Alvarez TL. From convergence insufficiency to functional reorganization: A longitudinal randomized controlled trial of treatment-induced connectivity plasticity. CNS Neurosci Ther. 2024 Aug;30(8):e70007. doi: 10.1111/cns.70007. PMID 39185637
- [Derived] Hajebrahimi F, Gohel S, Scheiman M, Sangoi A, Iring-Sanchez S, Morales C, Santos EM, Alvarez TL. Altered Large-Scale Resting-State Functional Network Connectivity in Convergence Insufficiency Young Adults Compared With Binocularly Normal Controls. Invest Ophthalmol Vis Sci. 2023 Nov 1;64(14):29. doi: 10.1167/iovs.64.14.29. PMID 37982763
- [Derived] Alvarez TL, Scheiman M, Morales C, Gohel S, Sangoi A, Santos EM, Yaramothu C, d'Antonio-Bertagnolli JV, Li X, Biswal BB. Underlying neurological mechanisms associated with symptomatic convergence insufficiency. Sci Rep. 2021 Mar 22;11(1):6545. doi: 10.1038/s41598-021-86171-9. PMID 33753864
- [Derived] Alvarez TL, Scheiman M, Santos EM, Morales C, Yaramothu C, D'Antonio-Bertagnolli JV, Biswal BB, Gohel S, Li X. The Convergence Insufficiency Neuro-mechanism in Adult Population Study (CINAPS) Randomized Clinical Trial: Design, Methods, and Clinical Data. Ophthalmic Epidemiol. 2020 Feb;27(1):52-72. doi: 10.1080/09286586.2019.1679192. Epub 2019 Oct 22. PMID 31640452